CLINICAL TRIAL: NCT04807543
Title: Effect of Progesterone on Latent Phase Prolongation in Patients With Preterm Premature Rupture of Membranes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ppprom
Record Dates: First submitted 2021-02-20; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Preterm Premature Rupture of Membrane
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — 17 alpha-Hydroxyprogesterone Caproate; Castor Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- study group (Active Comparator): 17-hydroxyprogesterone caproate (17P) (250 mg in castor oil, 1 mL total volume)intramuscular injection
  Interventions: Drug: 17-hydroxyprogesterone caproate
- control group (Placebo Comparator): castor oil, 1 mL total volume intramuscular injection
  Interventions: Drug: Castor Oil

INTERVENTIONS:
Drug: 17-hydroxyprogesterone caproate — intramuscular injection weekly
  Arms: study group
Drug: Castor Oil — intramuscular injection weekly
  Arms: control group

SUMMARY:
The aim of the study is to assess the efficacy of 17-hydroxyprogesterone caproate (17P) therapy on the latency period in pregnant women with Preterm premature rupture of membranes.

DETAILED DESCRIPTION:
After taking informed written consent, the recruited patients will be subjected to the following:

1. Detailed history

   * Personal History: Name, age ,residence ,special habits of medical importance
   * Obstetric history: first day of last menstrual period for accurate estimation of gestational age and antenatal care
   * Past history: history of any medical disorder or surgical history with particular emphasis on prior PPROM or preterm labor
   * History of the present pregnancy: Medical or surgical condition to define high risk pregnancy.
2. Examination of the patients General examination: blood pressure, pulse, temperature

   Abdominal examination:
   * Inspection: fundal level, scars, umbilicus.
   * Palpation: presence of contractions, fetal lie and presentation.
   * Pelvic Examination only by sterile speculum to exclude cord prolapse , bloody liquor and cervical dilatation and effacement
   * Non stress test to ensure reassuring fetal well being
   * Ultrasound examination to:-

     * Assess fetal viability.
     * Amniotic fluid index.
     * Determine gestational age.
     * Exclude major anomalies.
     * Placental location.
3. Baseline laboratory investigations:

   * Complete blood count (CBC).
   * Prothrombin time (PT).
   * Activated partial thromboplastin time (aPTT).
   * Liver and kidney function.

The included patients were randomized using sealed opaque envelope method into one of two groups:

Group I (study group): in which 17-hydroxyprogesterone caproate (17P) (250 mg in castor oil, 1 mL total volume, intramuscular injection weekly) will be administered.

Group II (control group): in which an identical-appearing placebo (1 mL castor oil only) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age between 24 and 34 weeks

Exclusion Criteria:

* Medical or obstetric conditions that could put them at risk for uterine atony , postpartum hemorrhage AND infection, such as

  * Emergency Cesarean section.
  * Chorioamnionitis.
  * Placenta previa.
  * Multiple gestation.
  * Preeclampsia.
  * Macrosomia.
* Non reassuring fetal status or fetal distress
* Presence of fetal anomalies incompatable with life
* Woman with antepartum haemorrhage
* Diagnosis of Established preterm labor

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
prolongation of the pregnancy until a favorable gestational age | 10 to 12 weeks (up to 34.0 weeks of gestation or documentation of fetal lung maturity at 32.0 to 33.9 weeks.)
  The most common method of measuring gestational age in weeks is by calculating the time since the last menstrual period based on dates provided by a woman at the first prenatal visit IF not available first trimester Ultrasound will be used

SECONDARY OUTCOMES:
Latency . | 10 to 12 weeks (interval in weeks from randomization to delivery)
  The most common method of measuring gestational age in weeks is by calculating the time since the last menstrual period based on dates provided by a woman at the first prenatal visit IF not available first trimester Ultrasound will be used
Composite neonatal morbidity | 1 week (from delivery to 1 week post Natal)
  by Apgar score ,blood gases ,and labs

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: starting 6 months after publication